CLINICAL TRIAL: NCT05568407
Title: A NIS of Avelumab in Real-World Treatment for Patients With Advanced or Metastatic Urothelial Cancer in Argentina and Brazil -LATAM AVENUE
Brief Title: A Study of Avelumab in Real-World Treatment for Patients With Advanced or Metastatic Urothelial Cancer
Status: Terminated | Type: Observational
Why Stopped: The trial terminated due to the inability to recruit the planned number of subjects. The decision was not based on any safety and/or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B9991050; LATAM AVENUE (Other: Alias Study Number)
Record Dates: First submitted 2022-09-23; First posted 2022-10-05 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — avelumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with Advanced or Metastatic Urothelial Cancer: Patients with Advanced or Metastatic Urothelial Cancer
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — As used in real world practice

SUMMARY:
This ambispective (both retrospective and prospective) NIS will evaluate the effectiveness and safety of Avelumab as a maintenance therapy administered after completion of first-line platinum-based chemotherapy in patients with locally advanced or metastatic urothelial cancer under routine conditions of daily clinical practice in Argentina and Brazil in line with the approved Avelumab label indication. Primary objective: • To evaluate overall survival (OS) rate at 12 and 24- months after the index date (date of the first Avelumab administration) in patients treated with Avelumab maintenance therapy. Secondary objectives: • To assess OS in patients treated with Avelumab maintenance therapy. To assess progression-free survival (PFS) of patients treated with Avelumab maintenance therapy. • To evaluate safety and tolerability of Avelumab maintenance therapy. • To assess duration of treatment (DOT) between the first and last dose of avelumab. • To describe the clinical and demographics characteristics of Argentinean and Brazilian patients treated with Avelumab maintenance therapy. Other objectives: • To evaluate anti-tumor effectiveness of Avelumab maintenance therapy.

DETAILED DESCRIPTION:
Urothelial carcinoma are tumors originating from the urothelial cells that line the bladder, renal pelvis, ureter, and urethra. Each year, bladder cancer (BC) accounts for 3.0% of global cancer diagnoses, with more than 570,000 new cases diagnosed and 2.1% of new deaths, with more than 210,000 deaths worldwide. In Latin America, BC placed the 10th and 9th positions in the incidence of cancer in Argentina and Brazil, respectively, and both countries have BC as the 5th most frequent cancers among males excluding non-melanoma skin cancer. 2-4 Among men, BC is the 6th most common cancer and the 9th leading cause of cancer death. Incidence and mortality in males are approximately four times higher compared to women with BC globally. In 2020, Argentina and Brazil reported over 3,700 and 15,800 new cases of BC, respectively. The 5-year prevalence at all ages of 11,401 (25 per 100,000) in Argentina and 43,545 (20 per 100,000) in Brazil. Besides male population, other risk factors for BC include prevalence of tobacco smoking, infection with Schistosoma haematobium, occupational exposures to organic solvents, and arsenic contamination in drinking water. 2,5 First-line standard of care for patients with advanced or metastatic urothelial cancer is a platinum-based chemotherapy regimen; however, the median OS in patients treated with Cisplatin-based chemotherapy is only 12-14 months, approximately. Besides, most patients with advanced or metastatic urothelial cancer commonly experience disease progression within 9 months after initiation of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, ≥18- years of age at the time of Avelumab treatment initiation
2. Patients with locally advanced or metastatic urothelial cancer with any histology (histologically confirmed, unresectable locally advanced or metastatic urothelial carcinoma and/or documented Stage IV disease (per American Joint Committee on Cancer/International Union for Cancer Control TNM system1 19-21) at the start of first-line chemotherapy)
3. Patients who have completed first-line platinum-based chemotherapy with no evidence of disease progression according to medical chart (ie, with a SD, PRor complete response [CR]).
4. Patients who are receiving or have received at least one dose of Avelumab as the firstl ine maintenance therapy according to label indication
5. Patients with ongoing treatment with Avelumab who provided written informed consent allowing the data collection. For decease patients and those who are lost to follow-up, an approved ICF waiver is allowed.

Exclusion Criteria:

* Patients who have participated in any interventional clinical trial of a drug or device within 28- days prior to the start of Avelumab maintenance therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Adult patients, ≥18- years of age at the time of Avelumab treatment initiation
  2. Patients with locally advanced or metastatic urothelial cancer with any histology (histologically confirmed, unresectable locally advanced or metastatic urothelial carcinoma and/or documented Stage IV disease (per American Joint Committee on Cancer/International Union for Cancer Control TNM system1 19-21) at the start of first-line chemotherapy)
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 36 months
  To evaluate OS rate at 12- and 24- months after the index date (date of the first Avelumab administration) in patients treated with Avelumab maintenance therapy.

SECONDARY OUTCOMES:
Progression-Free Survival | 36 months
  Patients treated with Avelumab maintenance therapy
OS | 36 months
  In patients treated with Avelumab maintenance therapy
Duration Of Treatment | 36 months
  Between the first and last dose of Avelumab
Frequency and nature of all-cause adverse events (AEs) | 36 months
  Toxicity; Dosage change (frequency and dosses approved); Progression disease; Cardiological Abnormalities; Dyspnea; Cough; Pneumonitis; Lab Abnormalities
Frequency of all-cause AEs leading to discontinuation or interruption of Avelumab maintenance therapy | 36 months
  Progression disease; Toxicity; Patient Decision
Duration of Avelumab maintenance therapy among the patients who discontinued the study drug due to all-cause AEs | 36 months
  Disease progression; Toxicity; Patient Decision
Frequency of potential signs and symptoms of immune-related AEs | 36 months
  Dyspnea; Fatigue; Rush; Glottis Edema; Cardiological Abnormalities; Cough; Pneumonitis
Frequency of patients with Avelumab dosing change due to any AE related to this drug | 36 months
  Dosage decrease for toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Argentina (3):
  - Alexander Fleming S.A (Instituto Medico Especializado Alexander Fleming), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Comite de Etica de la Investigacion del Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Sanatorio Privado de la Cañada, Córdoba
- Brazil (4):
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus/Aesc, Porto Alegre, Rio Grande do Sul
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Oncoclínicas Do Brasil Servicos Médicos S/A - Oncocentro, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991050